CLINICAL TRIAL: NCT01574378
Title: Cost Effectiveness and Clinical Outcomes of Wound Closure Using V-Loc™ 90 Sutures.
Brief Title: Effectiveness of Wound Closure Using V-Loc™ 90 Sutures in Lipoabdominoplasty Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vladimir Grigoryants MD (Other)
Responsible Party: Sponsor-Investigator, Vladimir Grigoryants MD, sponsor investigator, Grigoryants Medical Corporation
Organization: Grigoryants Medical Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: vl12345
Record Dates: First submitted 2011-11-28; First posted 2012-04-10 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Open Surgical Wounds
Keywords: Abdominoplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm (Active Comparator): Control arm- conventional method of wound closure
  Interventions: Device: conventional closure
- V-Loc group (Experimental): V-Loc 90 barbed sutures
  Interventions: Device: V-Loc 90

INTERVENTIONS:
Device: conventional closure — non barbed sutures used to close wounds Conventional three layer wound closure using non-locking sutures polyglactin 910 (Vicryl, Ethicon) and polyglecaprone 25 (Monocryl, Ethicon)
  Arms: Control arm
Device: V-Loc 90 — 2-layer wound closure using V-Loc 90 barbed suture
  Arms: V-Loc group

SUMMARY:
VLock suture studied in abdominal wound closure. Time and cosmesis was studied

ELIGIBILITY:
Inclusion Criteria:

* lipoabdominoplasty patients

Exclusion Criteria:

* poor health,
* history of radiation,
* smoking

Ages: 32 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
closure time | 1 day
  operative closure time studied

SECONDARY OUTCOMES:
Safety- number of complications | 12 months
  Number of complications on control incisions vs number of complications on experimental incisions
Cosmesis | 12 months
  Scar thickness and appearance

CONTACTS AND LOCATIONS:
Locations (1):
- Vladimir Grigoryants, MD, Glendale, California, United States